CLINICAL TRIAL: NCT02267044
Title: Effective Pain Management of Continuous Versus Single Shot Injection Interscalene Block During Shoulder Replacement Surgery
Brief Title: Effective Pain Management of Interscalene Blocks During Shoulder Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14061
Record Dates: First submitted 2014-08-12; First posted 2014-10-17 (Estimated); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Primary Osteoarthritis, Unspecified Shoulder
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ropivacaine Single Shot Block (Active Comparator): Single Shot Interscalene block patients will receive a single shot of 30ml of 0.5% Ropivacaine prior to surgery
  Interventions: Drug: Ropivacaine
- Ropivacaine Continuous block (Active Comparator): Continuous Interscalene block patients will receive a shot of up to 30ml of 0.5% Ropivacaine and then a catheter is placed. The catheter is secured with Dermabond and Tegaderm. Once surgery is complete, the catheter is connected to a pain ball system which holds 400ml of 0.2% Ropivacaine local anesthetic. The rate is locked in at 8ml/hr. Catheter is pulled once the pain ball is empty.
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — The drug used for the interscalene blocks
  Other Names: Naropin

SUMMARY:
Shoulder replacement surgery is recognized as having the potential to cause a considerable amount of postoperative pain. Adequate management of pain after surgery is necessary not only to improve the patient's wellbeing but also to facilitate recovery. Several regional anesthesia techniques are available to combat postoperative pain in the shoulder replacement surgery patient, however, which method provides superior pain relief remains unknown. The purpose of this study is to examine the effectiveness of a continuous interscalene block versus a single shot interscalene block for postoperative pain relief in the shoulder replacement patient.

Patients undergoing shoulder replacement surgery will experience more effective pain relief with a continuous interscalene block versus and single shot interscalene block.

DETAILED DESCRIPTION:
This is a prospective randomized controlled trial. 76 patients receiving either primary total shoulder replacement, hemiarthroplasty, or reverse total shoulder replacement will be randomized to a regional anesthesia technique as part of their surgical procedure. 38 patients will receive a single shot interscalene block containing ropivicaine and 38 patients will receive a continuous interscalene block containing ropivicaine.

ELIGIBILITY:
Inclusion Criteria:

* Surgical candidate for primary total shoulder replacement, hemiarthroplasty, or reverse total shoulder replacement
* patient must be 18 years or older and willing to sign and date an Institutional Review Board informed consent form, and
* must be able to understand and agree to follow study protocol.

Exclusion Criteria:

* severe bronchopulmonary disease,
* oxygen dependent,
* existing nerve injury,
* BMI > 40,
* coagulation disorders,
* allergy to ropivicaine,
* history of drug or alcohol abuse,
* American Academy of Anaesthesiologists physical status classification > lll,
* pregnant women.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2014-08; Primary Completion 2016-10 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Pain Score Measure | participants will be followed for the duration of the hospital stay, an expected average of 3 days
  Patients will be assessed for pain levels by visual analog scale while in the hospital per nursing protocol. Electronic Medical Record will be used to acquire pain scores.

SECONDARY OUTCOMES:
Morphine Sulfate Equivalence consumption | participants morphine sulfate consumption will be gathered for the duration of the hospital stay, an expected average of 3 days
  Total Morphine Sulfate equivalence consumption for each post-operative day while in the hospital will be collected through Electronic medical record.
Pain control Satisfaction Score | 10 day post operative
  Patient's post operative pain control satisfaction score will be obtained at the first post operative follow up visit with the physician which is expected to occur on avearage 10 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Samer Hasan, MD, Principal Investigator — Cincinnati Sportsmedicine and Orthopaedic Center; Robert Rolf, MD, Principal Investigator — Beacon Orthopaedic Center
Locations (1):
- Good Samaritan Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Borgeat A, Tewes E, Biasca N, Gerber C. Patient-controlled interscalene analgesia with ropivacaine after major shoulder surgery: PCIA vs PCA. Br J Anaesth. 1998 Oct;81(4):603-5. doi: 10.1093/bja/81.4.603. PMID 9924240